CLINICAL TRIAL: NCT07239115
Title: Perioperative Randomized Evaluation of leVetiracetam's Efficacy and Safety for Epilepsy Prevention in Neurosurgical Tumor Patients (PREVENT): A Multicenter, Randomized, Double-Blind, Placebo-Controlled Parallel Trial
Brief Title: Levetiracetam for Seizure Prevention After Brain Tumor Surgery
Acronym: PREVENT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Wang Jia, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY2025-213-02
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Seizures After Brain Tumor Surgery
Keywords: Levetiracetam; Perioperative prophylaxis; Postoperative seizures; Tumor-related epilepsy; Antiseizure medication; PREVENT trial
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levetiracetam group (Experimental): Participants receive levetiracetam 500 mg intravenously 1 hour before surgery and again on the evening after surgery (around 20:00-22:00), followed by oral levetiracetam 0.5 g twice daily from postoperative day 2 through 3 months. Intravenous infusion is given over approximately 15 minutes after dilution in 100 mL 0.9% sodium chloride or 5% glucose.
  Interventions: Drug: Levetiracetam
- Placebo group (Placebo Comparator): Participants receive matching placebo solution intravenously 1 hour before surgery and again on the evening after surgery (around 20:00-22:00), followed by oral placebo tablets twice daily from postoperative day 2 through 3 months. The placebo is identical in appearance, packaging, and administration schedule to levetiracetam.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam 500 mg (5 mL) for intravenous infusion administered 1 hour before surgery and again on the evening after surgery (approximately 20:00-22:00), diluted in 100 mL 0.9% sodium chloride or 5% glucose and infused over about 15 minutes. From postoperative day 2 through 3 months, oral levetiracetam tablets 0.5 g twice daily (or via nasogastric route if oral intake not feasible) are administered.
  Arms: Levetiracetam group
Drug: Placebo — Matching placebo solution (5 mL) for intravenous infusion 1 hour before surgery and again on the evening after surgery (approximately 20:00-22:00), diluted in 100 mL 0.9% sodium chloride or 5% glucose and infused over about 15 minutes. From postoperative day 2 through 3 months, matching placebo tablets are given twice daily (oral or via nasogastric route). Placebo formulation, packaging, and administration schedule are identical to those of levetiracetam.
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the efficacy and safety of levetiracetam for the prevention of postoperative seizures in adult patients undergoing supratentorial brain tumor surgery. It is a multicenter, randomized, double-blind, placebo-controlled, parallel-group clinical trial. Eligible participants will be randomly assigned in a 1:1 ratio to receive levetiracetam or placebo, starting 1 hour before surgery and continuing for 3 months postoperatively. The primary outcome is the incidence of clinical seizures within 3 months after surgery. Secondary outcomes include subclinical seizures within 7 days and 3 months postoperatively, adverse events within 3 months, and health economic outcomes. The study aims to clarify the role of levetiracetam in the primary prevention of perioperative seizures in brain tumor patients and to provide evidence for rational use of antiseizure medications in neurosurgical practice.

DETAILED DESCRIPTION:
Seizures are a common complication in brain tumor patients, particularly after supratentorial craniotomy, with approximately two-thirds occurring within the first postoperative month and affecting both early recovery and long-term outcomes. Although prophylactic ASMs are widely used in practice, there is no consensus on whether routine prophylaxis is necessary or on the optimal regimen. Major societies generally conclude that evidence is insufficient to recommend for or against routine use, while some national guidance provides conditional suggestions only for "high-risk" patients-highlighting the lack of robust data. Real-world studies also show high but heterogeneous use and no unified standard. A high-quality randomized trial is therefore required to determine the necessity, efficacy, and safety of routine prophylaxis.

The PREVENT trial is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy and safety of levetiracetam in adults undergoing supratentorial tumor resection without a prior seizure history, and thereby to assess the need for routine perioperative prophylaxis. Participants are randomized 1:1 with center-stratified block allocation. The dosing regimen is: one intravenous dose 1 hour preoperatively and another on the evening after surgery, followed by oral/NG maintenance (0.5 g twice daily) through postoperative month 3; the control arm receives matching placebo. Standard antiseizure treatment is provided if seizures occur and these events are recorded as endpoints. Scheduled assessments occur at screening, day of surgery, postoperative day 7, month 3 (±7 days), and month 6 (±10 days).

The primary endpoint is clinical seizures within 3 months after surgery, adjudicated by predefined criteria. Secondary endpoints are subclinical seizures within 7 days and 3 months (based on standardized EEG review). Exploratory endpoints include direct medical costs and direct non-medical/indirect costs at 3 months, and clinical seizures within 6 months. Safety endpoints include adverse events, serious adverse events, and death through 3 months. The principal null hypothesis is no difference between groups. Efficacy is analyzed primarily in the full analysis set (FAS) with per-protocol (PPS) as supportive; center effects are modeled, two-sided α=0.05, and results reported as risk differences with 95% CIs and relative risks. The planned sample size is 558 participants across ~10 centers, with independent safety oversight. This trial will provide robust randomized evidence on the necessity, benefits, risks, and economic impact of routine perioperative prophylaxis to guide standardized clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing craniotomy for supratentorial brain tumor resection.
2. Radiologically confirmed supratentorial brain tumor (excluding posterior fossa tumor, brainstem tumor, or gliomatosis cerebri).
3. Age between 18 and 75 years.
4. No history of seizures or epilepsy.
5. No prior use of antiepileptic drugs.
6. Karnofsky Performance Status (KPS) score ≥ 70.
7. Signed written informed consent

Exclusion Criteria:

1. Concomitant brain injury (such as cerebrovascular accident, severe head trauma) or any intracranial disease other than tumor.
2. Pregnant or lactating women.
3. Intestinal stoma, cardiac disease, previous craniotomy for brain tumor resection, or intracranial infection.
4. Severe hepatic or renal dysfunction (defined as ALT or AST >3× upper limit of normal; serum creatinine >3.0 mg/dL [265.2 μmol/L] or eGFR <30 mL/min/1.73m²).
5. Significant electrolyte imbalance (severe hyponatremia: serum sodium <125 mmol/L; severe hypernatremia: serum sodium >160 mmol/L; severe hypocalcemia: serum calcium <2.5 mmol/L; or severe hypercalcemia: serum calcium >6.5 mmol/L).
6. Long-term history of psychiatric disorders, alcoholism, or drug abuse.
7. Severe mental illness.
8. Allergy to or contraindication for antiepileptic drugs.
9. Unable to undergo MRI or EEG examination.
10. Deemed unsuitable for participation by the investigator.
11. Participation in another drug or device clinical trial within the past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative clinical seizures within 90 days after surgery | Within 90 days after surgery
  The occurrence of one or more postoperative clinical seizures within 90 days after supratentorial brain tumor resection, confirmed by treating physicians and reviewed by independent neurologists. A clinical seizure is defined as a transient occurrence of signs or symptoms resulting from abnormal excessive or synchronous neuronal activity in the brain, with or without electrographic correlation. Seizure episodes will be classified according to the International League Against Epilepsy (ILAE) 2017 operational classification

SECONDARY OUTCOMES:
Incidence of postoperative subclinical seizures detected by EEG | Within 7 days and 3 months after surgery
  Occurrence of subclinical epileptiform discharges or electrographic seizures detected by scalp EEG within 7 days and 3 months postoperatively, without clinical seizure manifestations. Recordings will be reviewed and confirmed by independent neurophysiologists.
Safety outcomes: incidence of adverse events, serious adverse events, and all-cause mortality within 3 months after surgery | Within 3 months after surgery
  Composite safety outcomes include the proportion of participants experiencing any adverse events (AEs), serious adverse events (SAEs), or all-cause mortality within 3 months postoperatively. AEs and SAEs will be coded using MedDRA and evaluated for severity and relationship to study drug according to ICH-GCP definitions.

OTHER OUTCOMES:
Economic outcomes: direct medical, direct non-medical, and indirect costs within 3 months after surgery | Within 3 months after surgery
  Total healthcare and non-healthcare costs within 3 months postoperatively, including direct medical costs (hospitalization, surgery, medications), direct non-medical costs (transportation, accommodation), and indirect costs (loss of productivity, caregiver burden). Data will be collected from hospital billing systems and structured questionnaires.
Incidence of postoperative clinical seizures within 6 months after surgery | Within 6 months after surgery
  The proportion of participants experiencing one or more clinical seizures within 6 months after surgery, confirmed by investigators and reviewed by independent neurologists.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Dr.Jia, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China